CLINICAL TRIAL: NCT04210661
Title: Spelling Mistake Tolerant Word Prediction for Working, Writing and Communicating - Predict4All
Brief Title: Spelling Mistake Tolerant Word Prediction for Working, Writing and Communicating
Acronym: Predict4All
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A01882-55
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Dysorthographia; Neurologic Disorder
Keywords: word prediction; dysorthographia
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: interventionnal, prsopective, randomized, multicentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic prediction software (Active Comparator): test with classic precition software
  Interventions: Other: prediction software with spell checker
- prediction software with spell checker (Experimental): test with prediction software with spell checker
  Interventions: Other: prediction software with spell checker

INTERVENTIONS:
Other: prediction software with spell checker — test with prediction software with spell checker

SUMMARY:
The main objective of the PREDICT4ALL project is to provide written communication in a computer, reducing the number of spelling errors for each user.

The effectiveness of written communication is defined in this study by the number of spelling errors for each user. Word prediction (and therefore correction) must be able to be configured by a therapist (speech therapist, occupational therapist).

Adapting the prediction to user errors should also allow it to be more relevant throughout the text input. This software efficiency must increase text input speed, Reduce the cognitive load, establish a classification of spelling errors adapted to the context of text input speed and develop the word prediction module tolerant of these spelling errors.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 25 years old For center 1
* patient with dysorthographia
* educational level greater than or equal to CE2
* A developmental level in reading on the Evalouette test (Evaleo battery) greater than or equal to CE1 For center 2
* Neurologic disorder impacting communication

Exclusion Criteria:

* Patient's refusal to participate in the study
* Persons under guardianship
* Pregnant women
* No affiliation to a social security scheme (beneficiary or beneficiary)
* Having visual disturbances preventing the use of the computer tool

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
number of spelling errors | 20 min
  total of number of spelling errors during the test

SECONDARY OUTCOMES:
Text input speed | 20 min
  Text input speed in the test
Prediction usage rate | 20 min
  number of times the prediction is used
Keystrokes Saving Rate | 5 min
  measured by the percentage of input saved by word prediction versus a keyboard alone
Attentional load | 1 min
  Likert Analog Visual Scale [0-10]
Fatigue | 1 min
  Likert Analog Visual Scale [0-10]
software Satisfaction | 1 min
  Likert Analog Visual Scale [0-10]

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Raymond Poincaré hospital, Garches
  - CMRRF Kerpape, Ploemeur

IPD SHARING:
Plan to Share IPD: No